CLINICAL TRIAL: NCT01185808
Title: Vitamin D Supplementation in Chronic Rhinosinusitis With Nasal Polyps
Acronym: VDinCRS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Rodney J. Schlosser, PI, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vitamin D in CRSwNP
Record Dates: First submitted 2010-07-30; First posted 2010-08-20 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Chronic Sinusitis
Keywords: sinusitis; chronic sinusitis with polyps
MeSH Terms: conditions — Sinusitis | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Active Comparator): Vitamin D 5,000IU/day for 6 weeks
  Interventions: Biological: Vitamin D
- Placebo (Placebo Comparator): Placebo for 6 weeks.
  Interventions: Biological: Vitamin D

INTERVENTIONS:
Biological: Vitamin D — Vitamin D 5000IU/day for 6 weeks
  Other Names: Vitamin D3

SUMMARY:
The purpose of this study is to determine if Vitamin D supplementation improves clinical and immunologic parameters in chronic rhinosinusitis with nasal polyps.

DETAILED DESCRIPTION:
Introductory Statement: Our laboratory has found that patients with chronic rhinosinusitis with nasal polyps (CRSwNP) have insufficient levels of vitamin D3. This is a proposal to conduct a placebo controlled trial on the use of vitamin D3 (5,000IU/day for 6 weeks) to determine clinical and immunologic outcomes in these patients.

General Investigational Plan: We routinely examine vitamin D levels in all patients with CRSwNP. Those that are insufficient (less than 32 ng/ml) and have agreed to undergo sinus surgery will be randomized to placebo or vitamin D3 supplementation (5,000IU/day) for 6 weeks prior to surgery. Blood will be drawn pre- and post-supplementation to examine systemic immune parameters such as dendritic cell and T cell expression and cytokine levels. Sinus tissue will be collected at the time of surgery to analyze local immune parameters (dendritic cell, T cell and cytokine levels) between supplemented and placebo groups. Clinical outcomes will be analyzed using quality of life questionnaires, endoscopic grading and nasal peak inspiratory flow pre- and post- supplementation. IRB approval for this research project is pending.

ELIGIBILITY:
Inclusion Criteria:

* Chronic sinusitis with polyps

Exclusion Criteria:

* Use of systemic steroids, or other immunmodulatory agents in preceding monthS, other immunologic, renal, gastrointestinal, endocrine or skeletal disorder (rheumatoid arthritis, immunodeficiency, cystic fibrosis, ciliary dyskinesia, malabsorption, etc.)
* Pregnancy or age less than 14 years.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Clinical symptom score | 6 weeks
  Symptoms will be graded using Sinonasal Outcomes Test-22.

SECONDARY OUTCOMES:
Nasal peak inspiratory flow | 6 weeks
  Measurement of maximal nasal peak inspiratory flow
Systemic and local immunologic parameters | 6 weeks
  Histologic analysis of sinus immune cells, as well as systemic measurement of immune cells.

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Schlosser, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States